CLINICAL TRIAL: NCT00765388
Title: A Comparative, Randomised, Crossover Study With 2 Urostomy Bags Among 30 Urostomy-operated Persons in UK
Brief Title: A Randomised Cross-over Study With Two 1-piece Urostomy Bags.
Acronym: DK188OS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DK188OS
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2012-08

CONDITIONS: Urostomy
Keywords: urostomy, 1-piece, cross-over, randomised, preference

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SenSura Uro (Experimental): The test product is a CE-marked non-sterile one-piece urostomy multi-chamber bag with the SenSura adhesive.
  Interventions: Device: SenSura Uro
- hollister Uro (Active Comparator): The comparator product is CE-marked and non-sterile and produced for urostomy operated. It is a flat one-piece urostomy product, Hollister Moderma Flex Urostomy beige, Cut-to-Fit Bag, flat adhesive
  Interventions: Device: Hollister

INTERVENTIONS:
Device: SenSura Uro — The test product is a CE-marked non-sterile one-piece urostomy multi-chamber bag with the SenSura adhesive.
  Other Names: SenSura URO Standard Wear 1-piece bag; Product number:1438298
  Arms: SenSura Uro
Device: Hollister — The comparator product is CE-marked and non-sterile and produced for urostomy operated. It is a flat one-piece urostomy product, Hollister Moderma Flex Urostomy beige, Cut-to-Fit Bag, flat adhesive.
  Other Names: Moderma Flex Urostomy, Cut-to-fit bag, flat adhesive.; product id : 29100
  Arms: hollister Uro

SUMMARY:
Background Urostomy is a surgical procedure that detours or diverts urine away form a diseased or defective bladder. The bladder can be removed and the urine is passed out of the body through an opening (stoma) in the stomach. People with urostomy will not be able to start and stop urine coming out through the stoma, so a urostomy bag will be fitted to collect the urine as it comes out.

A urostomy bag consists of an adhesive, which is attached to the skin around the stoma and a bag connected to the adhesive to collect the urine.

It is very important the standard is high on these products; otherwise the user (urostomy-patient) will experience lots of problems with the skin around the stoma.

DETAILED DESCRIPTION:
In this trial we are comparing two types of urostomy bags - the SenSura 1-piece and Hollisters Moderma Flex.

Both products are CE-marked, meaning that they are safe and approved in use for people with an urostomy.

Population 30 urostomy operated people from UK will participate in the trial. Only participants who normally use a flat 1-piece urostomy bag can participate. It is very important that the participants keep their normal use- and change pattern. Furthermore they need to be over 18 years old, have had the urostomy for more than 3 months, the size of the urostomy shall be between 15-55 mm, otherwise the bag will not fit them and then they should be able to handle the bags themselves and be willing to use the two products tested in the trial.

ELIGIBILITY:
Inclusion Criteria:

In order to be enrolled in the clinical investigation, the subject must:

* Be at least 18 years old,
* Be mentally and physically capable of signing the written consent form
* Be able to fill in the Case Report Form (questionnaire)
* Have an urostomy with a size between 15-55 mm.
* Have had the urostomy for 3 months or more,
* Use a 1-piece bag normally.
* Be able to handle the bag themselves (application and removal)
* Be willing to use Coloplast SenSura 1-piece bag
* Be willing to use Hollisters Moderma Flex, 1-piece bag

Exclusion Criteria:

In order to be enrolled in the clinical investigation, the subjects must not:

* Be a convex base plate user (i.e. a bowl-shaped adhesive which pushes the stoma forward)
* Need to use an ostomy belt
* Be currently suffering from any dermatologiacal problems, needing special treatment, in the peristomal area (investigator will evaluate skin according to a newly developed ostomy skin tool from Coloplast A/S)
* Being treated with chemo- or radiation therapy,
* Be hospitalized during study enrollment, or have a hospitalization or significant surgery planned during the 4-week study period, or
* Be pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Katte, Stoma Nurse, Study Chair — Ashford and St. Peters Hospital; Maureen Bridgland, Stoma Nurse, Principal Investigator — Royal Sussex County Hospital; Caroline Rudoni, Stoma Nurse, Principal Investigator — St. Georges Hospital; Theresa Bowles, Stoma Nurse, Principal Investigator — Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK); Michael Lynch, Surgeon, Principal Investigator — Colchester General Hospital; Sharon Fillingham, Nurse, Principal Investigator — UCLH
Locations (6):
- United Kingdom (6):
  - St. Peters Hospital, Chertsey, Surrey
  - Caroline Rudoni, London, Tooting
  - Maureen Bridgland, Brighton
  - Michael Lynch, Colchester
  - University of London Hospital, London
  - Theresa Bowles, Norwich

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects where recruited by 6 stoma care sites in UK
Pre-assignment Details: No pre-assignment details
Groups:
- Hollister Uro First, Then SenSura Uro; SenSura Uro First, Then Hollister Uro: SenSura Uro (test product) and Hollister Uro (comparator) are CE-marked, non-sterile, 1-piece urostomy devices.
Period: Period 1
Arm/Group | Hollister Uro First, Then SenSura Uro | SenSura Uro First, Then Hollister Uro
Started | 16 (A cross-over study) | 11
Completed | 15 | 6
Not Completed | 1 | 5
Not completed — Lack of Efficacy | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Herpes Zoster | 0 | 1
Not completed — Hip operation | 0 | 1
Period: Period 2
Arm/Group | Hollister Uro First, Then SenSura Uro | SenSura Uro First, Then Hollister Uro
Started | 15 | 6
Completed | 15 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive SenSura Uro first and Hollister Uro first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 18
Region of Enrollment [Number; unit: participants]
  United Kingdom | 27

OUTCOME MEASURES:

1. Primary Outcome: Preference of Sensura vs Moderma
Description: Subjects were asked which of the tested products they preferred; SenSura or Moderma.
Time Frame: 4 weeks
Measure: Number; unit: percentage of prefering the product
Groups:
- SenSura Uro; Hollister Uro: SenSura Uro (test product)and Hollister Uro (comparator) are CE-marked, non-sterile, 1-piece urostomy devices.
Arm/Group | SenSura Uro | Hollister Uro
Number analyzed (Participants) | 27 | 27
percentage of prefering the product | 45 | 43

2. Secondary Outcome: Immediate Adhesion
Description: Evaluation of immediate adhesion after each period
Time Frame: 4 weeks
Population: Intention to treat (ITT)
Measure: Number; unit: Participants
Arm/Group | SenSura Uro | Hollister Uro
Number analyzed (Participants) | 21 | 20
Participants
  Very poor | 1 | 1
  Poor | 1 | 4
  Reasonable | 8 | 4
  Good | 7 | 6
  Very good | 4 | 5
Statistical Analysis 1: Comparison: SenSura Uro vs Hollister Uro; Test type: Superiority or Other; p = 0.96, Regression, Logistic; An ordinal logistic regression model. The null hypothesis tested is that there is no difference in the multinomial distributions defined by products

3. Secondary Outcome: Removal of the Bag
Description: How easy/difficult it was to remove the bag
Time Frame: 4 weeks
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | SenSura Uro | Hollister Uro
Number analyzed (Participants) | 22 | 23
Participants
  Very easy | 5 | 5
  Easy | 12 | 11
  Reasonable | 5 | 7
  Difficult | 0 | 0
  Very difficult | 0 | 0

4. Secondary Outcome: Adhesion of the Bag During Use
Description: Evaluation of the adhesion of the base plate around the stoma during use
Time Frame: 4 weeks
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | SenSura Uro | Hollister Uro
Number analyzed (Participants) | 22 | 23
Participants
  Very poor | 2 | 3
  Poor | 5 | 5
  Reasonable | 7 | 5
  Good | 3 | 6
  Very good | 5 | 4
Statistical Analysis 1: Comparison: SenSura Uro vs Hollister Uro; Test type: Superiority or Other; p = 0.92, Regression, Logistic; [statistical method as in outcome 2, analysis 1]

5. Secondary Outcome: Adhesives Ability to Absorb Perspiration
Description: Evaluation of the adhesives ability to absorb perspiration from the skin
Time Frame: 4 weeks
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | SenSura Uro | Hollister Uro
Number analyzed (Participants) | 21 | 22
Participants
  Very poor | 1 | 0
  Poor | 2 | 4
  Reasonable | 8 | 7
  Good | 6 | 9
  Very good | 4 | 2

6. Secondary Outcome: Flexibility of the Product
Description: Evaluation of the ability of the bag to conform with the patients movements (flexibility)
Time Frame: 4 weeks
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | SenSura Uro | Hollister Uro
Number analyzed (Participants) | 22 | 23
Participants
  Very poor | 1 | 1
  Poor | 0 | 4
  Reasonable | 8 | 5
  Good | 8 | 10
  Very good | 5 | 3
Statistical Analysis 1: Comparison: SenSura Uro vs Hollister Uro; Test type: Superiority or Other; p = 0.40, Regression, Logistic; An ordinal logistic regression model. The null hypothesis tested is that there is no difference inthe multinomial distributions defined by products

7. Secondary Outcome: Awareness of the Presence of the Product
Description: Evaluates the patients awareness of the presence of the product during use.
Time Frame: 4 weeks
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | SenSura Uro | Hollister Uro
Number analyzed (Participants) | 22 | 23
Participants
  Very much | 0 | 2
  Much | 1 | 3
  Some | 8 | 5
  A little | 11 | 10
  Not at all | 2 | 3
Statistical Analysis 1: Comparison: SenSura Uro vs Hollister Uro; Test type: Superiority or Other; p = 0.64, Regression, Logistic; [statistical method as in outcome 6, analysis 1]

8. Secondary Outcome: Feeling of Security During the Day
Description: The patients feeling of security with the bag during the day
Time Frame: 4 weeks
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | SenSura Uro | Hollister Uro
Number analyzed (Participants) | 22 | 23
Participants
  Very poor | 3 | 4
  Poor | 3 | 4
  Reasonable | 5 | 5
  Good | 7 | 7
  Very good | 4 | 3
Statistical Analysis 1: Comparison: SenSura Uro vs Hollister Uro; Test type: Superiority or Other; p = 0.55, Regression, Logistic; [statistical method as in outcome 6, analysis 1]

9. Secondary Outcome: Feeling of Security During the Night
Description: The patients feeling of security with the product during the night
Time Frame: 4 weeks
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | SenSura Uro | Hollister Uro
Number analyzed (Participants) | 22 | 23
Participants
  Very poor | 3 | 3
  Poor | 4 | 4
  Reasonable | 3 | 6
  Good | 6 | 7
  Very good | 6 | 3
Statistical Analysis 1: Comparison: SenSura Uro vs Hollister Uro; Test type: Superiority or Other; p = 0.48, Regression, Logistic; [statistical method as in outcome 6, analysis 1]

10. Secondary Outcome: Problems With Splashing Sounds During Use
Description: The patient was asked whether he/she noticed any splashinh sounds during use
Time Frame: 4 weeks
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | SenSura Uro | Hollister Uro
Number analyzed (Participants) | 22 | 23
Participants
  Very much | 0 | 1
  Much | 0 | 0
  Some | 3 | 3
  A little | 4 | 4
  Not at all | 15 | 15

11. Secondary Outcome: Bag Twisting During Night
Description: The patient was asked if he/she noticed whether the bag twisted during night
Time Frame: 4 weeks
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | SenSura Uro | Hollister Uro
Number analyzed (Participants) | 22 | 23
Participants
  Yes | 4 | 13
  No | 18 | 10

12. Secondary Outcome: Changes in Skin Compared to Before Study
Description: The patient was asked whether he/she experienced changes in the skin condition after testing the blue/red product
Time Frame: 4 weeks
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | SenSura Uro | Hollister Uro
Number analyzed (Participants) | 21 | 22
Participants
  No, it is the same | 17 | 19
  Yes, it is better | 0 | 1
  Yes, it is worse | 4 | 2

ADVERSE EVENTS:
Time Frame: AE data where collected from inclusion and till the two test periods where completed (maximum 34 days)
Groups:
- Hollister Uro; SenSura Uro: SenSura Uro (test product) and Hollister Uro (comparator) are CE-marked, non-sterile, 1-piece urostomy devices.
Arm/Group | Hollister Uro | SenSura Uro
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/11
Other Adverse Events (participants affected / at risk) | 0/16 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the Inventions subject to the prior written consent of Sponsor. The Investigator shall submit the manuscript to Sponsor for approval, provided however that the Investigator will submit the manuscript at least thirty (30) days before disclosure for such proposed publication. If Sponsor wishes to file patent applications on Inventions Sponsor is allowed to delay the publication upon to a maximum period of 6 months since he above-mentioned submission.